CLINICAL TRIAL: NCT00898911
Title: Prediction of Overall Survival Using Mass Spectrometry Profiling in Head and Neck Cancer Patients Treated With Epidermal Growth Factor Receptor Inhibitors
Brief Title: Blood Sample Analysis in Predicting Overall Survival in Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000600560; ECOG-E3301T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood sample analysis in predicting overall survival in patients with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To validate the mass spectrometry profile that is predictive of survival benefit in patients with recurrent or metastatic head and neck squamous cell carcinoma treated with EGFR inhibitors.

OUTLINE: Plasma and serum samples are analyzed by matrix-assisted laser desorption/ionization time-of-flight mass spectrometry and classified according to prognosis ("good" vs "poor") using a previously developed predictive algorithm.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent or metastatic head and neck squamous cell carcinoma
* Meets 1 of the following criteria:

  * Enrolled on clinical trial ECOG-E3301 and previously treated with irinotecan hydrochloride and docetaxel
  * Enrolled on clinical trial VU-VICC-HN-0501 and previously treated with docetaxel and bortezomib
* Plasma and serum samples available for analysis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E3301
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07-08 (Actual); Primary Completion 2012-04-08 (Actual); Study Completion 2012-04-08 (Actual)

PRIMARY OUTCOMES:
Overall survival measured in weeks | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, MD, Study Chair — Vanderbilt-Ingram Cancer Center